CLINICAL TRIAL: NCT03595124
Title: A Randomized Phase 2 Trial of Axitinib/Nivolumab Combination Therapy vs. Single Agent Nivolumab for the Treatment of TFE/Translocation Renal Cell Carcinoma (tRCC) Across All Age Groups
Brief Title: A Study to Compare Treatments for a Type of Kidney Cancer Called TFE/Translocation Renal Cell Carcinoma (tRCC)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2018-01489; NCI-2018-01489 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AREN1721 (Other: Children's Oncology Group); AREN1721 (Other: CTEP); U10CA180886 (NIH)
Record Dates: First submitted 2018-07-19; First posted 2018-07-23 (Actual); Results first posted 2025-10-10 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Renal Cell Carcinoma; Stage III Renal Cell Cancer AJCC v8; Stage IV Renal Cell Cancer AJCC v8; TFE3-Rearranged Renal Cell Carcinoma; Unresectable Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Axitinib; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A (axitinib, nivolumab) (Experimental): Patients receive axitinib PO BID on days 1-28 and nivolumab intravenously (IV) over 30 minutes, or per institutional guidelines, on days 1 and 15 (if < 18 years old) or on day 1 (if >= 18 years old). Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Axitinib; Biological: Nivolumab
- Arm B (axitinib) (Experimental): Patients receive axitinib PO BID on days 1-28. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. (CLOSED TO ACCRUAL AS OF 1/23/2020 - PROSPECTIVE PATIENTS ARE RANDOMLY ASSIGNED TO ARMS A OR C)
  Interventions: Drug: Axitinib
- Arm C (nivolumab) (Experimental): Patients receive nivolumab IV over 30 minutes, or per institutional guidelines, on days 1 and 15 (if < 18 years old) or on day 1 (if >= 18 years old). Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Drug: Axitinib — Given PO
  Other Names: AG 013736; AG-013736; AG013736; Inlyta
  Arms: Arm A (axitinib, nivolumab); Arm B (axitinib)
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm A (axitinib, nivolumab); Arm C (nivolumab)

SUMMARY:
This phase II trial studies how well axitinib and nivolumab work in treating patients with TFE/translocation renal cell carcinoma that cannot be removed by surgery (unresectable) or has spread to other places in the body (metastatic). Axitinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving axitinib and nivolumab may work better in treating patients with TFE/translocation renal cell carcinoma compared to standard treatment, including surgery, chemotherapy, or immunotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish the clinical activity, assessed primarily by progression-free survival, of nivolumab therapy with or without axitinib for advanced transcription factor E3/translocation morphology renal cell carcinoma (TFE/tRCC).

SECONDARY OBJECTIVE:

I. To further define the toxicities of the study arms in the treatment of translocation morphology RCC across all ages.

EXPLORATORY OBJECTIVES:

I. To characterize tRCC clinical behavior across all age groups. II. To evaluate type of antitumor immune response and stability of T cell activation before and after treatment with immunotherapy or antiangiogenic therapy.

III. To develop a tumor bank of tRCC tumor samples treated on study for further biological investigations.

IV. To characterize the pharmacokinetics of axitinib when given in combination with nivolumab in pediatric patients with tRCC.

OUTLINE: Patients are now randomized to 1 of 2 arms - Arm A or Arm C.

ARM A: Patients receive axitinib orally (PO) twice daily (BID) on days 1-28 and nivolumab intravenously (IV) over 30 minutes, or per institutional guidelines, on days 1 and 15 (if < 18 years old) or on day 1 (if >= 18 years old). Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive axitinib PO BID on days 1-28. Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity. (CLOSED TO ACCRUAL AS OF 1/23/2020 - PROSPECTIVE PATIENTS ARE RANDOMLY ASSIGNED TO ARMS A OR C)

ARM C: Patients receive nivolumab IV over 30 minutes, or per institutional guidelines, on days 1 and 15 (if < 18 years old) or on day 1 (if >= 18 years old). Treatment repeats every 28 days for up to 26 cycles (2 years) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 1 year, every 4 months for 1 year, and every 6 months for 2 years. Follow-up at year 5 and beyond is at the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >= 12 months at enrollment
* Patients must have a body surface area (BSA) >= 0.53 m^2
* Histologically confirmed unresectable or metastatic translocation morphology renal cell carcinoma diagnosed using World Health Organization (WHO)-defined criteria. Patients may be newly diagnosed or have received prior cancer therapy

  * Patients must have had histologic verification of the malignancy
  * Patients must have measurable disease, documented by clinical, radiographic, or histologic criteria as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1
  * Patients must have a tumor showing the appropriate morphologic appearance, and either confirmed TFE3 nuclear protein expression by immunohistochemistry with appropriate positive and negative controls performed at a Clinical Laboratory Improvement Act (CLIA)-certified laboratory, or evidence of TFE3 or TFEb translocation by either fluorescence in situ hybridization (FISH) or reverse transcriptase- polymerase chain reaction (RT-PCR) performed at a CLIA-certified laboratory. For TFE3 immunohistochemistry, any nuclear positivity in the presence of appropriate positive and negative controls should be considered as evidence of TFE3 immunohistochemical expression. NOTE: If the institution is unable to perform these studies, unstained slides may be submitted to Dr. Elizabeth Perlman, who will perform TFE3 analysis at no charge. The slide will be returned to the referring institution for local evaluation, to be included in their institutional report
* Patients must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients =< 16 years of age
* Patients must have a life expectancy of >= 8 weeks
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study

  * Myelosuppressive chemotherapy: Must not have received within 2 weeks of entry onto this study (6 weeks if prior nitrosourea)
  * Immunotherapy: Must not have received within 4 weeks of entry onto this study
  * Biologic (anti-neoplastic agent): At least 7 days since the completion of therapy with a biologic agent
  * Radiation therapy (RT): >= 2 weeks for local palliative RT (small port); >= 6 months must have elapsed if prior craniospinal RT or if >= 50% radiation of pelvis; >= 6 weeks must have elapsed if other substantial bone marrow (BM) radiation
* Peripheral absolute neutrophil count (ANC) >= 1000/uL (performed within 7 days prior to enrollment)
* Platelet count >= 75,000/uL (transfusion independent) (performed within 7 days prior to enrollment)
* Hemoglobin >= 8.0 g/dL (may receive red blood cell [RBC] transfusions) (performed within 7 days prior to enrollment)
* Urine protein: =< 30 mg/dL in urinalysis or =< 1+ on dipstick, unless quantitative protein is < 1000 mg in a 24 hours (h) urine sample (performed within 7 days prior to enrollment)
* For patients < 18 years of age: Serum creatinine =< 1.5 x upper limit of normal (ULN), or measured or calculated creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 for patient with creatinine levels > 1.5 x institutional ULN, or a serum creatinine based on age/gender as follows (performed within 7 days prior to enrollment):

  * 1 to < 2 years - 0.6 mg/dL (male, female)
  * 2 to < 6 years - 0.8 mg/dL (male, female)
  * 6 to < 10 years - 1 mg/dL (male, female)
  * 10 to < 13 years - 1.2 mg/dL (male, female)
  * 13 to < 16 years - 1.5 mg/dL (male), 1.4 mg/dL (female)
  * >= 16 years - 1.7 mg/dL (male), 1.4 mg/dL (female)
  * Creatinine clearance should be calculated per institutional standard
* For patients >= 18 years of age: Serum creatinine =< 2 x ULN, or measured or calculated creatinine clearance or radioisotope GFR >= 40 mL/min/1.73 m^2 for patient with creatinine levels > 2 x institutional ULN (performed within 7 days prior to enrollment)

  * Creatinine clearance should be calculated per institutional standard
* Serum total bilirubin =< 1.5 x ULN for age, or direct bilirubin =< ULN for patients with total bilirubin levels > 1.5 X ULN (performed within 7 days prior to enrollment)
* Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) < 3 x ULN for age (performed within 7 days prior to enrollment)
* Albumin > 2.5 mg/dL (performed within 7 days prior to enrollment)
* Shortening fraction of >= 27% by echocardiogram, or
* Ejection fraction of >= 50% by radionuclide angiogram
* No history of myocardial infarction, severe or unstable angina, or peripheral vascular disease
* Corrected QT (QTc) =< 480 msec. Note: Patients with grade 1 prolonged QTc (450-480 msec) at the time of study enrollment should have correctable causes of prolonged QTc addressed if possible (i.e., electrolytes, medications)
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN. However, if patient is receiving anticoagulant therapy, PT or partial thromboplastin time (PTT) should be within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless patient is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* A baseline blood pressure (BP) =< the 95th percentile for age, height, and gender for patients < 18 years old, or =< 150 mmHg (systolic) and =< 90 mmHg (diastolic) for patients >= 18 years old

  * Note: 2 serial blood pressures should be taken at least 1 hour apart and averaged to determine baseline BP
* Patients are eligible if on stable doses (>= 7 days) of anti-hypertensive medications with a baseline BP meeting the criteria above

Exclusion Criteria:

* Patients unable to swallow whole tablets
* Patients who in the opinion of the investigator are not able to comply with the study procedures are not eligible
* Prior Therapy

  * Patients who have received prior therapy with axitinib, nivolumab, or other PD1/PD-L1 targeted therapies
  * Patients who have received prior therapy with more than one anti VEGF based agent (antibody or tyrosine kinase inhibitor)
  * Patients with hypersensitivity to axitinib, nivolumab, or any of its excipients
  * Patients who previously received an allogeneic stem cell transplant (SCT) or solid organ transplant are not eligible
  * Patients may not be receiving any other investigational agents (within 4 weeks prior to study enrollment)
  * Patients who have received prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study enrollment or who have not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks prior to enrollment
  * Surgery: Patients who have had or who are planning to have the following invasive procedures are not eligible:

    * Major surgical procedure, laparoscopic procedure, open biopsy, core biopsy, fine needle aspirate, or significant traumatic injury within 7 days prior to enrollment. NOTE: External central lines must be placed at least 3 days prior to planned treatment initiation and subcutaneous ports must be placed at least 7 days prior to planned treatment initiation
    * Patients who are planning cytoreductive surgery within the first 12 weeks following therapy initiation
    * Patients who have a serious or non-healing wound or ulcer at the time of study enrollment are not eligible
  * Patients who have a history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 28 days of study enrollment are not eligible
  * Patients who have received prior targeted small molecule therapy within 2 weeks of enrollment or have not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks prior to enrollment. NOTE: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Pre-existing conditions, which may include:

  * Additional known malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer
  * Patients with underlying immune deficiency, chronic infections including hepatitis, tuberculosis (TB), or autoimmune disease
  * Human immunodeficiency virus (HIV)-infected patients with the exception of patients on an effective anti-retroviral therapy with an undetectable viral load within 6 months prior to enrollment
  * Patients with underlying hematologic issues including congenital bleeding diathesis, known previous gastrointestinal (GI) bleeding requiring intervention within the past 6 months, history of hemoptysis within 42 days prior to study enrollment, active pulmonary emboli, or deep vein thromboses (DVT) that are not stable on anticoagulation regimen
  * Patients must not have had significant vascular disease (i.e. Moya-Moya, aortic aneurysm requiring surgical repair)
  * A known history of, or any evidence of active, non-infectious pneumonitis
  * Patients with known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease. Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to study enrollment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to study enrollment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
  * Any uncontrolled, intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
  * Any serious medical or psychiatric illness/condition including substance use disorders likely in the judgment of the investigator(s) to interfere or limit compliance with study requirements/treatment
  * Patients with active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Treatments and/or medications the patient is receiving or has received that would make her/him ineligible, including:

  * Concomitant (or receipt of) treatment with medications that may affect the metabolism of nivolumab and/or axitinib within 7 days prior to planned first dose of protocol therapy
  * A live vaccine within 30 days of planned first dose of protocol therapy. NOTE: Inactivated flu vaccines are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Pregnancy and breast feeding

  * Due to risks of fetal and teratogenic adverse events as seen in animal studies, a negative pregnancy test must be obtained in females of childbearing potential, defined as females who are post-menarchal. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * Females of childbearing potential that are sexually active must agree to either practice 2 medically accepted highly-effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 5 months after the last dose of study drug
  * Lactating females are not eligible unless they have agreed not to breastfeed their infants starting with the first dose of study therapy through 5 months after the last dose of study therapy
* Male patients of reproductive potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy. Prior history of vasectomy does not replace requirement for contraceptive use
* Regulatory requirements

  * All patients and/or their parents or legal guardians must sign a written informed consent
  * All institutional, Food and Drug Administration (FDA), and National Cancer Institute (NCI) requirements for human studies must be met

Min Age: 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2026-11-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James I Geller, Principal Investigator — Children's Oncology Group
Locations (269):
- United States (268):
  - Children's Hospital of Alabama, Birmingham, Alabama
  - CTCA at Western Regional Medical Center, Goodyear, Arizona
  - Cancer Center at Saint Joseph's, Phoenix, Arizona
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - Mission Hope Medical Oncology - Arroyo Grande, Arroyo Grande, California
  - PCR Oncology, Arroyo Grande, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Mercy Cancer Center - Carmichael, Carmichael, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Kaiser Permanente Downey Medical Center, Downey, California
  - Mercy Cancer Center - Elk Grove, Elk Grove, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Mattel Children's Hospital UCLA, Los Angeles, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Mercy Cancer Center - Rocklin, Rocklin, California
  - Mercy Cancer Center - Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Pacific Central Coast Health Center-San Luis Obispo, San Luis Obispo, California
  - Mission Hope Medical Oncology - Santa Maria, Santa Maria, California
  - Woodland Memorial Hospital, Woodland, California
  - Children's Hospital Colorado, Aurora, Colorado
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Saint Francis Cancer Center, Colorado Springs, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rocky Mountain Hospital for Children-Presbyterian Saint Luke's Medical Center, Denver, Colorado
  - CommonSpirit Cancer Center Mercy, Durango, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - AdventHealth Littleton, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - AdventHealth Parker, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Golisano Children's Hospital of Southwest Florida, Fort Myers, Florida
  - UF Health Cancer Institute - Gainesville, Gainesville, Florida
  - Nemours Children's Clinic-Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - Nemours Children's Hospital, Orlando, Florida
  - Saint Joseph's Hospital/Children's Hospital-Tampa, Tampa, Florida
  - Saint Mary's Medical Center, West Palm Beach, Florida
  - Children's Healthcare of Atlanta - Arthur M Blank Hospital, Atlanta, Georgia
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Saint Jude Midwest Affiliate, Peoria, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Riley Hospital for Children, Indianapolis, Indiana
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - UI Health Care Mission Cancer and Blood - West Des Moines Clinic, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Laurel Clinic, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Saint Joseph Hospital, Lexington, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Saint Joseph London, London, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Norton Children's Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - UofL Health Medical Center Northeast, Louisville, Kentucky
  - Saint Joseph Mount Sterling, Mount Sterling, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Henry Ford Health Saint John Hospital, Detroit, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Minnesota Oncology - Burnsville, Burnsville, Minnesota
  - Cambridge Medical Center, Cambridge, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Clinics and Surgery Center Maple Grove, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - Monticello Cancer Center, Monticello, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - Fairview Northland Medical Center, Princeton, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Cardinal Glennon Children's Medical Center, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Nebraska Cancer Specialists/Oncology Hematology West PC, Grand Island, Nebraska
  - Fred and Pamela Buffett Cancer Center - Kearney, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - Las Vegas Urology - Green Valley, Henderson, Nevada
  - Oncology Las Vegas - Henderson, Henderson, Nevada
  - Urology Specialists of Nevada - Green Valley, Henderson, Nevada
  - Desert West Surgery, Las Vegas, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Hope Cancer Care of Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - Urology Specialists of Nevada - Central, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Las Vegas Urology - Sunset, Las Vegas, Nevada
  - Urology Specialists of Nevada - Southwest, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Oncology Las Vegas - Tenaya, Las Vegas, Nevada
  - OptumCare Cancer Care at MountainView, Las Vegas, Nevada
  - Urology Specialists of Nevada - Northwest, Las Vegas, Nevada
  - Alliance for Childhood Diseases/Cure 4 the Kids Foundation, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Town Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Cancer Care Specialists - Reno, Reno, Nevada
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Albany Medical Center, Albany, New York
  - Maimonides Medical Center, Brooklyn, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - NYP/Columbia University Medical Center/Herbert Irving Comprehensive Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Mission Hospital, Asheville, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's Hospital, Dayton, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - ProMedica Toledo Hospital/Russell J Ebeid Children's Hospital, Toledo, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Treatment Centers of America, Tulsa, Oklahoma
  - Legacy Emanuel Children's Hospital, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Prisma Health Cancer Institute - Spartanburg, Boiling Springs, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Cancer Institute - Laurens, Clinton, South Carolina
  - Prisma Health Cancer Institute - Easley, Easley, South Carolina
  - Prisma Health Cancer Institute - Butternut, Greenville, South Carolina
  - Prisma Health Cancer Institute - Faris, Greenville, South Carolina
  - Prisma Health Cancer Institute - Eastside, Greenville, South Carolina
  - Prisma Health Cancer Institute - Greer, Greer, South Carolina
  - Prisma Health Cancer Institute - Seneca, Seneca, South Carolina
  - Memorial Hospital, Chattanooga, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - Saint Jude Children's Research Hospital, Memphis, Tennessee
  - The Children's Hospital at TriStar Centennial, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Dell Children's Medical Center of Central Texas, Austin, Texas
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - El Paso Children's Hospital, El Paso, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Children's Hospital of San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - University Hospital, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Hospital, Salt Lake City, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Children's Hospital of The King's Daughters, Norfolk, Virginia
  - Overlake Medical Center, Bellevue, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Saint Michael Cancer Center, Silverdale, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Mary Bridge Children's Hospital and Health Center, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Holy Family Memorial Hospital, Manitowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Marinette, Marinette, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - HSHS Saint Nicholas Hospital, Sheboygan, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
- HIMA San Pablo Oncologic Hospital, Caguas, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A (Axitinib, Nivolumab) | Arm B (Axitinib) | Arm C (Nivolumab)
Started | 7 | 3 | 5
Completed | 1 | 0 | 0
Not Completed | 6 | 3 | 5
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Ineligible | 1 | 1 | 0
Not completed — Disease Progression | 4 | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Axitinib, Nivolumab) | Arm B (Axitinib) | Arm C (Nivolumab) | Total
Number analyzed (Participants) | 7 | 3 | 5 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 1 | 4 | 10
  Between 18 and 65 years | 2 | 2 | 1 | 5
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.7 (8.2) | 21.5 (5.9) | 18.4 (13.6) | 18.2 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 1 | 4
  Male | 4 | 3 | 4 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 0 | 4
  Not Hispanic or Latino | 4 | 2 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 2
  White | 4 | 1 | 2 | 7
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 2 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 7 | 3 | 5 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: The Kaplan-Meier method will be used to estimate 1-year PFS, defined as the time from randomization to disease progression or death due to any cause. The 70% confidence interval was chosen to match the one-sided significance level of alpha = 0.15 specified in the protocol analysis plan.
Time Frame: Up to 1 year from study entry
Population: The data was analyzed with revised intention-to-treat approach. The following patients were excluded: Three (3) Arm B patients (as of Amendment 2A, the arm permanently closed to accrual and patients were randomly assigned to Arms A and C), One (1) Arm A patient who is ineligible for the study. 11 total patients were analyzed.
Measure: Number (70% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Axitinib, Nivolumab) | Arm C (Nivolumab)
Number analyzed (Participants) | 6 | 5
percentage of participants | 33 [18.32 to 60.64] | 0 [NA to NA] — All Arm C patients experienced progression

2. Secondary Outcome: Overall Survival (OS)
Description: The Kaplan-Meier method will be used to estimate 1-year OS, defined as the time from study entry until death. The 70% confidence interval was chosen to match the one-sided significance level of alpha = 0.15 specified in the protocol analysis plan.
Time Frame: Up to 1 year from study entry
Population: as for outcome 1
Measure: Number (70% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Axitinib, Nivolumab) | Arm C (Nivolumab)
Number analyzed (Participants) | 6 | 5
percentage of participants | 100 [NA to NA] — Zero Arm A patients experienced death | 80 [63.45 to 100]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: The ORR will be defined as the proportion of patients that achieve a complete or partial response according to RECIST version 1.1 among patients who initiated protocol therapy and completed at least one subsequent imaging assessment. The 70% confidence interval was chosen to match the one-sided significance level of alpha = 0.15 specified in the protocol analysis plan.
Time Frame: Up to 1 year from study entry
Population: as for outcome 1
Measure: Number (70% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Axitinib, Nivolumab) | Arm C (Nivolumab)
Number analyzed (Participants) | 6 | 5
percentage of participants | 33 [11.50 to 62.18] | 0 [0 to 31.54]

4. Secondary Outcome: Percentage of Patients Experiencing Adverse Events (AEs)
Description: Percentage of patients experiencing grade 3+ non-hematologic and all grade 4-5 AEs occurring during protocol therapy or within 30 days of treatment will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. The 70% confidence interval was chosen to match the one-sided significance level of alpha = 0.15 specified in the protocol analysis plan.
Time Frame: Up to 2 years from study entry
Population: as for outcome 1
Measure: Number (70% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A (Axitinib, Nivolumab) | Arm C (Nivolumab)
Number analyzed (Participants) | 6 | 5
percentage of participants | 50 [30.52 to 69.48] | 80 [46.87 to 97.39]

5. Other Pre Specified Outcome: Translocation Morphology Renal Cell Carcinoma Clinical Behavior
Description: Site(s) of disease at presentation (including extent of lymph node involvement), site(s) of relapse, surgical and radiotherapy practices on protocol therapy.
Time Frame: Up to 2 years from study entry
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Type of Antitumor Immune Response and Stability of T Cell Activation
Description: Levels of protocol-specified marker analytes and tumor expression before and after treatment and changes due to treatment will be described using descriptive statistics.
Time Frame: Up to 1 year from study entry
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Pharmacokinetics (PK) Parameters of Axitinib
Description: PKs will be evaluated at day 1 of cycles 1, 2, and 3.
Time Frame: Up to 12 weeks from study entry
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 5 years after randomization
Description: Adverse event reporting is collected routinely using case report forms. The SAE table reflects NCI Common Terminology Criteria for Adverse Events (CTCAEs) submitted by the institution via expedited reporting (NCI AdEERs / CAeRs). All remaining CTCAEs collected by means other than expedited reporting are non-serious and are reported in the "AE Other" table. All-Cause Mortality includes all deaths collected on the study. Ineligible patients are excluded from reporting of adverse events.
Arm/Group | Arm A (Axitinib, Nivolumab) | Arm B (Axitinib) | Arm C (Nivolumab)
All-Cause Mortality (participants affected / at risk) | 1/6 | 2/2 | 4/5
Serious Adverse Events (participants affected / at risk) | 4/6 | 2/2 | 5/5
Other Adverse Events (participants affected / at risk) | 2/6 | 0/2 | 1/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Axitinib, Nivolumab) (N=6) | Arm B (Axitinib) (N=2) | Arm C (Nivolumab) (N=5)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Chylous ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Disease progression (General disorders) | 0 (0) | 2 (2) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
subcutaneous perianal abscess (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Axitinib, Nivolumab) (N=6) | Arm B (Axitinib) (N=2) | Arm C (Nivolumab) (N=5)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (4) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (5) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Decreased T4 (Investigations) | 1 (1) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Elevated Platelets (Investigations) | 1 (1) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (3) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (5) | 0 (0) | 0 (0)
Hemoglobin increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (6) | 0 (0) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (7) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroid stimulating hormone increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
acne (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03595124/Prot_SAP_000.pdf
  • Informed Consent Form: PAREN1721_A09Consent(Untracked).pdf (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03595124/ICF_001.pdf
  • Informed Consent Form: PAREN1721_A09Consent2(Untracked).pdf (2021-12-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT03595124/ICF_002.pdf